CLINICAL TRIAL: NCT06086899
Title: The Effect of Early MSAT Treatment on Radiating Pain in the Upper Extremity Caused by Traffic Accidents: A Pragmatic Randomized Controlled Trial
Brief Title: The Efficacy and Safety of Early MSAT on Radiating Pain in the Upper Extremity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JS-CT-2023-06
Record Dates: First submitted 2023-10-12; First posted 2023-10-17 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Radiating Pain in the Upper Extremity
Keywords: Motion Style Acupuncture Treatment; Radiating pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: A Pragmatic randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cervical motion style acupuncture treatment(Trapezius, Rhomboid, Scalene) (Experimental): The MSAT group recieved 3 sessions of MSAT; on second, third, fourth day after hospitalization. A trained doctor of Korean medicine with at least 3 years of clinical experience conducted the MSAT.
  The MSAT group were also treated with other Korean medical treatment everyday: acupuncture, chuna, pharmacoacupuncture and Korean herbal medicine.
  Interventions: Procedure: Cervical motion style acupuncture treatment(Trapezius, Rhomboid, Scalene); Procedure: Korean medical treatment
- Korean medical treatment (Active Comparator): The control group were received Korean medical treatment everyday after hospitalization: acupuncture, chuna, pharmacoacupuncture and Korean herbal medicine.
  Interventions: Procedure: Korean medical treatment

INTERVENTIONS:
Procedure: Cervical motion style acupuncture treatment(Trapezius, Rhomboid, Scalene) — Motion Style Acupuncture Treatment(MSAT) is a therapeutic technique using acupuncture needle created in Jaseng Hospital. This treatment involves patients with musculoskeletal pain to move the part of their body actively during acupuncture treatment under physicians' observation
  Arms: Cervical motion style acupuncture treatment(Trapezius, Rhomboid, Scalene)
Procedure: Korean medical treatment — acupuncture treatment, chuna, pharmacoacupuncture, Korean herbal medicine

SUMMARY:
This study is a double blind, randomized controlled trail. condition/disease: radiating pain in the upper extremity. treatment/intervention: motion style acupuncture treatment

DETAILED DESCRIPTION:
"Motion Style Acupuncture Treatment(MSAT) is a therapeutic technique using acupuncture needle created in Jaseng Hospital. This treatment involves patients with musculoskeletal pain to move the part of their body actively during acupuncture treatment under physicians' observation. This treatment is known to relieve the pain and increase the range of motion(ROM). However, there has been no specific value for the effect of this treatment.

So, we conducted a randomized controlled trials to verify the efficacy and safety of MSAT on radiating pain in the upper extremity. From October 2023 to December 2024, we collected 100 inpatients who were suffered from radiating pain in the upper extremity with the numeric rating scale(NRS) over 5 after injury by acute traffic accident(TA). For experimental group(n=50), we conducted MSAT three times(on 2nd, 3rd and 4th day of hospitalization) and other Korean medical treatment. For control group(n=50), just Korean medical treatment except MSAT was conducted. For these two groups, we compared NRS, Visual Analogue Scale(VAS), Neck Disability Index(NDI), C-SPINE MRI, EuroQol 5-Dimension (EQ-5D) and Patient Global Impression of Change (PGIC)."

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 19-69 years on the date they sign the consent form.
* Patients who are suffered byradiating pain in the upper extremity that occurred within 3 days after traffic accident.
* Patients who are hospitalized due to traffic accident.
* Patients with NRS of radiating pain ≥ 5.
* Patients who provide consent to participate in the trial and return the informed consent form.

Exclusion Criteria:

* Patients with a specific serious disease that may cause radiating pain: malignancy, spondylitis, inflammatory spondylitis, etc.
* Patients with progressive neurological deficits or with severe neurological symptoms.
* Patients with medical history of cervical surgery or thoracic surgery within the last three weeks.
* Patients who have radiating pain in upper extremity before the traffic accident.
* Patients with a specific serious disease that may interfere with the interpretation of the therapeutic effects or results: malignancy, spondylitis, inflammatory spondylitis, etc.
* Patients who are taking steroids, immunosuppressants, mental illness drugs, or other drugs that may affect the results of the study.
* If acupuncture is inadequate or unsafe: patients with hemorrhagic, receiving anticoagulants, severe diabetes and cardiovascular disease.
* Patients who are pregnant or planning to become pregnant.
* Patients who are participated in clinical trials other than observational studies without therapeutic intervention.
* Patients who are difficult to complete the research participation agreement.
* Other patients whose participation in the trial is judged by a researcher to be problematic.

Ages: 19 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-11-06 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale(NRS) of radiating pain | Screening, Baseline(day2), day3, day4, day5, Discharge 1 day, 1month after enrollment, 3month after enrollment
  NRS is a pain scale in which the patient indicates their subjective pain as a whole number from 0 to 10. The participant is asked to report their leg pain and discomfort using NRS, where 0 indicates 'no pain or discomfort' and 10 indicates 'the most severe pain and discomfort imaginable'.

SECONDARY OUTCOMES:
Location of Radiating pain | Baseline(day2), day3, day4, day5, Discharge 1 day, 1month after enrollment, 3month after enrollment
  The location of radiating pain varies depending on the nerve. The assessor will ask patients where the pain occur.
VAS of Radiating pain | Baseline(day2), day3, day4, day5, Discharge 1 day, 1month after enrollment, 3month after enrollment
  VAS is an assessment index in which the patient records their pain on a 100mm line from 'no pain' at one end, and 'the most severe pain imaginable' at the other end.
C-SPINE MRI | Taken within ±14 days of hospitalization
  We will examine the results of patients who underwent MRI. The investor will conduct whether or not MRI was performed, date of operation, presence of cervical disc herniation, grade of cervical disc herniation, area of cervical disc herniation, classification of disc degeneration, presence of stenosis.
NRS of Neck pain | Baseline(day2), day3, day4, day5, Discharge 1 day, 1month after enrollment, 3month after enrollment
  NRS is a pain scale in which the patient indicates their subjective pain as a whole number from 0 to 10. The participant is asked to report their leg pain and discomfort using NRS, where 0 indicates 'no pain or discomfort' and 10 indicates 'the most severe pain and discomfort imaginable'.
NDI | Baseline(day2), day5, Discharge 1 day, 1month after enrollment, 3month after enrollment
  NRS is a pain scale in which the patient indicates their subjective pain as a whole number from 0 to 10. The participant is asked to report their leg pain and discomfort using NRS, where 0 indicates 'no pain or discomfort' and 10 indicates 'the most severe pain and discomfort imaginable'.
EQ-5D | Baseline(day2), day5, Discharge 1 day, 1month after enrollment, 3 months after enrollment
  The EQ-5D is a method of indirectly calculating the weights of certain health states for quality of life after a multidimensional investigation of health states, and is the most widely used instrument for this purpose. The EQ-5D consists of 5 questions about current health state (mobility, self-care, usual activities, pain, anxiety/depression), and each question is scored on a 5-point Likert scale (1=no problems, 3=moderate problems, 5=severe problems). In this study, the investigators will use the Korean version of the EQ-5D, which has been demonstrated to be valid.
PGIC | day5, Discharge 1 day, 1month after enrollment, 3 months after enrollment
  The PGIC is an index that assesses improvements in functional limitation caused by whiplash injury. Participants rate the improvement in functional limitations after treatment on a 7-point Likert scale (1=Very much improved, 4=No change, 7=Very much worse). This index was originally developed for use in Psychology, but is currently used in various other medical fields to assess improvements in pain

CONTACTS AND LOCATIONS:
Overall Officials: In-Hyuk Ha, phD, Principal Investigator — Jaseng Medical Foundation
Locations (1):
- Jaseng Hospital of Korean Medicine, Seoul, Gangnam-Gu, South Korea

IPD SHARING:
Plan to Share IPD: No